CLINICAL TRIAL: NCT03281434
Title: The Effects of Whey Versus Collagen Protein Intake on Acute and Longer-term Skeletal Muscle Protein Synthesis in Older Adults
Brief Title: The Effects of Whey vs. Collagen on MPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HIREB 3916
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Aging
Keywords: Skeletal muscle; Protein synthesis; Protein ingestion; Resistance exercise

STUDY DESIGN:
Intervention Model Description: Parallel group design (with repeated measurements within each group)
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen peptide (Active Comparator): Supplement will be delivered twice daily (30g per supplement) of hydrolyzed collagen peptides
  Interventions: Dietary Supplement: Collagen peptide
- Whey protein (Experimental): Supplement will be delivered twice daily (30g per supplement) of whey protein isolate
  Interventions: Dietary Supplement: Whey protein isolate

INTERVENTIONS:
Dietary Supplement: Collagen peptide — Low leucine content protein supplement to be consumed twice daily
  Arms: Collagen peptide
Dietary Supplement: Whey protein isolate — High quality protein (DIAAS score), high leucine supplement, to be consumed twice daily
  Arms: Whey protein

SUMMARY:
With aging there is a natural loss of muscle mass and strength called sarcopenia, which increases the risk of falls and metabolic disease (i.e. Type II diabetes) and decreases the ability to perform activities of daily living. Eating protein and doing resistance exercise both increase the body's ability to make muscle protein, which is important to offset losses in muscle mass; however, older adults have a lower appetite and do not consume enough calories or protein to crease muscle and as such investigations in this population are needed. The amino acid (the building blocks of proteins) leucine is known to increase the ability of protein to make muscle. In this study we will investigate the ability of beverages with different types of protein and leucine to create muscle in older men and women whoa re particularly vulnerable to muscle losses and do not eat enough protein and are understudied in this area.

DETAILED DESCRIPTION:
The age-related decline in skeletal muscle mass and strength, termed sarcopenia, is associated with a host of metabolic disease states including, but not limited to, cancer, stroke, microvascular disease, type 2 diabetes, Parkinson's and Alzheimer's. Moreover, declines in skeletal muscle mass also are accompanied by an even more precipitous reduction in skeletal muscle strength, known as dynapenia, which is a predisposition for disability and falls. Sarcopenia begins in the 5th decade of life and proceeds, at least based on population-derived estimates, at a ~0.8% loss annually, with strength losses being greater and more variable at 2-5% year past the age of 50. Strategies to offset the loss of muscle mass with aging are imperative for the maintenance of quality of life and ability to perform activities of daily living in an older population.

Losses of skeletal muscle mass are underpinned by an imbalance between rates of muscle protein synthesis (MPS) and muscle protein breakdown (MPB). In healthy humans it is known that the change in the rate of MPS in response to contractile activity and protein feeding is the primary locus of control for human muscle mass. With aging, basal levels of MPS do not change in comparison to younger adults, however elevation in MPS response following an anabolic stimulus such as resistance exercise or protein ingestion are blunted when participants are exposed to the same stimulus, termed anabolic resistance. For example, older adults require 3-6 times the amount of resistance exercise volume and a 0.4 g/kg compared to 0.24 g/kg dose of high quality protein into order to stimulate basal rates of muscle protein synthesis.

Protein quality and dose are also critical when targeting maximal increases in MPS. The importance of amino acid digestibility is crucial as undigested dietary proteins may be unabsorbed and excreted rather than being absorbed in the small intestine or contributions to lean mass. The Food and Agriculture Organization has endorsed the digestible indispensable amino acid score (DIAAS) to assess protein quality as it is able to distinguish between proteins that were previously classed at an equivalent value. Using the DIAAS, proteins with the highest digestibility and quality scores are the two main milk proteins casein and whey, which have scores of 1.18 and 1.09, respectively whereas hydrolyzed collagen peptides (derived from bones and cartilaginous tissues) has a score of 0 as it lacks the amino acid tryptophan. Importantly, casein and whey have higher leucine contents than collagen peptides, including more of other essential amino acids. This is particularly important as data from our own laboratory has demonstrated that increasing the leucine concentration of a low protein mixed macronutrient beverage rescues rates of postprandial MPS to those seen with higher protein content. Moreover, leucine is a key trigger of the mechanistic target of rapamycin complex 1 (mTORC1), a 280-kDa serine/threonine kinase known to activate key translation initiation factors involved in MPS. Thus, protein doses of lower quality such as hydrolyzed collagen would in theory require a greater dose in order to elicit a similar response to whey or casein.

The use of hydrolyzed collagen as a supplement to enhance skeletal muscle anabolism has been scarcely examined previously literature with most studies in humans involving the use of collagen peptide supplementation to enhance collagen-containing tissues such as hair, skin and cartilaginous joints. Of the current literature, supplementation with collagen peptides in combination with resistance exercise was found to have remarkable effects on the accrual of lean mass in older men with a concomitant remarkable decrease in fat mass within a 12-week training period. It was also found to have remarkable effects on nitrogen balance in older women in comparison to whey protein despite a leucine content in collagen that is 1/16th of that found in whey protein isolate. If the anabolic potential of hydrolyzed collagen is able to match that of whey protein, it may provide an important, cost effective, and feasible method by which older adults are able to achieve suggested protein recommendations.

Protein ingestion following resistance exercise provides a potent and additive stimulus over either anabolic influence alone. A resistance exercise bout has been shown to sensitize the muscle to the effects of protein. Our lab has previously shown that older adults achieve the greatest increase in MPS following a resistance exercise bout when consuming 40 g of whey protein and that this effect was greater than consuming 40 g of protein without exercise. It will be crucial to our understanding of the protein needs of older adults to determine whether consumption of whey protein and collagen peptides are indeed equivalent and can be used to augment the muscle protein synthetic response following resistance exercise in older adults.

Many studies that assess acute changes in rates of MPS in response to protein intake do so by infusing a labeled amino acid tracer and calculating the incorporation of that tracer into skeletal muscle over a period of hours. While this approach provides important information, especially when coupled with quantitative measures of changes in muscle mass such a MRI, the assessment of tracer-infusion measured MPS is limited to ~5-6 h. Thus, recent developments of analytical techniques have enabled the use of a deuterated water methodology that enables assessment of MPS with much longer periods of incorporation i.e., days-to-weeks. Indeed, this method has been recently validated and its use is now becoming the interest of many researchers. However, only a few laboratories have demonstrated the ability to competently perform this measurement. In fact, we have recently conducted two studies using this methodology, and the MPS values that we obtained are entirely consistent with published reports. We propose that the use of the deuterated water methodology in combination with the use of stable isotope tracers, will provide us with measurements of MPS in both a controlled-acute and a free-living situation and would be a substantial advance in determining mechanisms underpinning protein ingestion and aging.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Ambulatory, and able to perform exercise
* Active (~3500-10,000 steps per day)

Exclusion Criteria:

* Smoker
* Diabetic
* Chronic conditions
* Consumption of medications known to affect muscle protein synthesis
* Statin myalgia
* Allergy to milk protein

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Acute myofibrillar muscle protein synthesis | 8 hours
  Assessed with stable isotope tracer infusion ([L-ring] 13C6 phenylalanine)
Medium length myofibrillar muscle protein synthesis | 7 days
  Assessed with deuterated water

SECONDARY OUTCOMES:
Fasted glucose, insulin and oxidative stress (IL6, TNF-a, CRP) | Assessed every 2 days throughout the 7 day monitoring period
  Measured with a fasted blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D., Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario
  - Ivor Wynne Center, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oikawa SY, Kamal MJ, Webb EK, McGlory C, Baker SK, Phillips SM. Whey protein but not collagen peptides stimulate acute and longer-term muscle protein synthesis with and without resistance exercise in healthy older women: a randomized controlled trial. Am J Clin Nutr. 2020 Mar 1;111(3):708-718. doi: 10.1093/ajcn/nqz332. PMID 31919527